CLINICAL TRIAL: NCT05862545
Title: Outcomes in Real-life After Initation Of treatmeNt With Trixeo (Budesonide / Glycopyrronium / Formoterol), a Non-interventional, Multi-centre, Prospective Cohort Study in Italian Routine Care Setting
Brief Title: Outcomes in Real-life After Initation of Treatment With Trixeo (Budesonide / Glycopyrronium / Formoterol)
Acronym: CHOROS ORION
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00076
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Disease, Chronic Obstructive, Patient Reported Outcome Measures
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Budesonide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients: Patients with COPD that start BGF treatment (The decision to prescribe BGF must be independent of enrolment into the study, must be determined by the treating physician and should be taken according to the standard of current best medical practice and national guideline)
  Interventions: Drug: BGF (budesonide/glycopyrrolate/formoterol fumarate)

INTERVENTIONS:
Drug: BGF (budesonide/glycopyrrolate/formoterol fumarate) — BGF is a maintenance treatment in adult patients with moderate to severe chronic obstructive pulmonary disease (COPD) who are not adequately treated by a combination of an ICS and a LABA, or a combination of a LABA and a LAMA. The decision to start treatment with BGF must be made by the treating physician according to the subjects' medical need and a positive benefit/risk balance. The decision to prescribe BGF must be independent of enrolment into the study, must be determined by the treating physician and should be taken according to the standard of current best medical practice and national guidelines.

SUMMARY:
The aim of the CHOROS ORION study is to describe patients' clinical and self-reported outcomes of treatment with BGF in Italy through effectiveness, clinical and self-reported measures assessed pre- and post-treatment initiation, up to one year of observation period. The study will focus primarily on the change in self-perceived health status in the first 12 weeks of treatment. This will allow to assess the short-term impact of treatment, thus contributing to fill the gap of knowledge from the current available medical literature. Moreover, in order to provide also a broader view, patients will be followed up to 52 weeks, where possible. The study results will be interpreted in the context of an observational study design where multiple factors, in addition to the new treatment, may contribute to the treatment effect.

DETAILED DESCRIPTION:
The therapeutic goal of chronic obstructive pulmonary disease (COPD) management is mainly reduction of symptoms and severity of exacerbations.Triple therapy (the combination of an ICS, a LABA and a LAMA) in a single fixed-dose combination is a valuable development in the treatment of COPD. On top of treatment adherence enhancement [Gaduzo et al., 2019], trials showed triple therapy improving lung function, Patients-Reported Outcomes (PROs), health-related quality of life, as well as lowering exacerbations and hospitalization rate compared to dual or mono-therapy [Bourbeau et al., 2021; Zheng et al, 2018].

Budesonide/glycopyrrolate/formoterol fumarate, hereafter BGF, is a maintenance treatment in adult patients with moderate to severe COPD who are not adequately treated by a combination of an ICS and a LABA, or a combination of a LABA and a LAMA. The availability of single-inhaler triple therapies in routine care may improve symptoms control, reduce exacerbation rate and COPD-related healthcare costs, thus leading to an improvement in patient health status and quality of life. However, real-world studies focusing on PROs are still limited.

The aim of the CHOROS ORION study is to describe patients' clinical and self-reported outcomes of treatment with BGF in Italy through effectiveness, clinical and self-reported measures assessed pre- and post-treatment initiation, up to one year of observation period. The study will focus primarily on the change in self-perceived health status in the first 12 weeks of treatment. This will allow to assess the short-term impact of treatment, thus contributing to fill the gap of knowledge from the current available medical literature. Moreover, in order to provide also a broader view, patients will be followed up to 52 weeks, where possible. The study results will be interpreted in the context of an observational study design where multiple factors, in addition to the new treatment, may contribute to the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged >= 40;
2. Physician-diagnosed COPD;
3. Signed written informed and privacy consent prior to study participation;
4. Patients starting treatment with BGF as prescribed according to the label, local market reimbursement criteria, and AIFA Nota 99;
5. Patients must be able and willing to read and to comprehend written instructions, and to comprehend and complete the questionnaires required by the protocol.

Exclusion Criteria:

1. COPD due to documented α-1 antitrypsin deficiency;
2. Patients with controlled COPD treated with triple fixed-dose combination in 12 months prior to screening visits;
3. Hospitalisation due to COPD exacerbation within the last 30 days prior to enrolment;
4. Pregnancy or lactation period;
5. Participation in a non-interventional observational trial that might, in the investigator's opinion, influence the assessment for the current study, or participation in any interventional, observational or clinical trial in the last 30 days prior to enrolment.

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with moderate to severe COPD who are eligible for BGF therapy, enrolled consecutively by physicians in specialist setting. The decision to start treatment with BGF must be made by the treating physician according to the subjects' medical need and a positive benefit/risk balance. The decision to prescribe BGF must be independent of enrolment into the study, must be determined by the treating physician and should be taken according to the standard of current best medical practice and national guidelines.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) score | baseline, 12 weeks after treatment start
  The change from baseline in COPD Assessment Test (CAT) score after 12 weeks treatment will be analysed using the within person difference between baseline and 12 weeks. Descriptive statistics (mean, median, standard deviation, interquartile range, minimum and maximum) will be provided. The mean change from baseline will be presented along with the 95% CI

SECONDARY OUTCOMES:
Baseline features | Baseline
  To describe the baseline features of patients starting BGF treatment in a real-world setting, in terms of demographics and clinical characteristics, COPD treatment paths and healthcare resource utilization in the previous year.
Impact of COPD on patients' life based on CAT | baseline, 26 and 52 weeks
  To describe the impact of COPD on patients' life, and how it changes over time during the observation period of treatment with BGF, administered as per routine clinical practice. COPD Assessment Test (CAT) questionnaire at baseline and after 26 and 52 weeks after BGF treatment start. In case of patient early withdrawal, CAT questionnaire will also be collected at the end of observation.
Patients' satisfaction to BGF | baseline, 26 and 52 weeks
  9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) at baseline, 26 and 52 weeks from treatment start. In case of patient early withdrawal, TSQM-9 questionnaire will also be collected at the end of observation.
Patient dyspnoea based on Modified Medical Research Council Dyspnoea Scale (mMRC) | Baseline, 26 and 52 weeks
  To describe patient dyspnoea and how it changes over time during the observation period of treatment with BGF, administered as per routine clinical practice. Modified Medical Research Council Dyspnoea Scale (mMRC) questionnaire at baseline, 26 and 52 weeks from treatment start. In case of patient early withdrawal, mMRC questionnaire will also be collected at the end of observation.
Eosinophil count | baseline, 26 and 52 weeks
  To describe the eosinophil count during the observation period of treatment with BGF, administered as per routine clinical practice. Eosinophil count in peripheral blood at baseline visit, and 26- and 52-week visits, which will occur after BGF treatment start, where available.
Responder Rate based on CAT | 12 weeks
  To describe the Responder Rate based on the CAT after 12 weeks of initiating treatment with BGF as per routine clinical practice. Number and rate of responders of the CAT [MID=2] after 12 weeks of BGF treatment.
Overall change in health status based on Patient Global Impression of Severity (PGIS) questionnaire | Baseline, 12, 26 and 52 weeks
  To assess patient-reported overall change in health status since the start of study treatment and overall global impression of severity during the observation period of treatment with BGF as per routine clinical practice. Single-item patient severity of COPD symptoms using PGIS at baseline, 12, 26 and 52 weeks after BGF treatment start. In case of patient early withdrawal, PGIS questionnaire will also be collected at the end of observation.
Exacerbation rate | 52 weeks
  To describe the occurrence of moderate - severe COPD exacerbations during the observation period of treatment with BGF, administered as per routine clinical practice. Number of moderate - severe COPD exacerbations, occurred during the BGF observation period and Annualized rate of moderate - severe COPD exacerbations during the BGF treatment observation period
Lung function | 52 weeks
  Describe Lung function parameters as measured at baseline and 52-week visit, available as per routine clinical practice.
OCS use | 52 weeks
  To describe the Oral Corticosteroids (OCS) use during the observation period of treatment with BGF, administered as per routine clinical practice, and in the previous year. OCS use during the observation period after BGF treatment start, and OCS use in the 52 weeks before BGF treatment start.
HCRU | 52 weeks
  To describe the healthcare resource utilization related to COPD during the observation period of treatment with BGF, administered as per routine clinical practice, and in the previous year. The number of GP/specialist visits, ER admissions, and hospitalizations (along with duration) related to COPD during the BGF observation period and the 52 weeks prior baseline will be described. The annualised rate of utilization per each type will be calculated.
Safety (frequency of all AEs, SAEs, AEs related to BGF and Special Situations during the observation period) | 52 weeks
  To describe safety profile of BGF during the observation period Absolute and relative frequency of all AEs, SAEs, AEs related to BGF and Special Situations during the observation period will be calculated. Moreover, the count of such events will be provided. Descriptive statistics will also be provided for severity, seriousness criteria (where applicable), relation grade with BGF, action taken and outcome.

OTHER OUTCOMES:
Relation between patient CAT score (dependent variable of interest) and patient baseline characteristics | 52 weeks
  To describe the relation of baseline characteristics and the impact of COPD on patients' life during the observation period of treatment with BGF, administered as per routine clinical practice
Baseline variables associated with exacerbations | 52 weeks
  To describe the relation of baseline characteristics and occurrence of COPD exacerbations during the observation period of treatment with BGF, administered as per routine clinical practice. The analysis will be performed in steps. Firstly, univariate Poisson regression models for the estimated impact on exacerbations occurrence during the observation period will be estimated independently considering the baseline variables (age, sex, BMI, smoking status, eosinophil count in peripheral blood, COPD phenotype and years from diagnosis, number of previous MACEs, number of moderate - severe COPD exacerbations in the year before BGF treatment start, and OCS use in the year before BGF treatment start). Then a multivariate Poisson regression model will be estimated including relevant variables (i.e. with a significant estimated coefficient), as evaluated through the single univariate regression models and the number of exacerbations during follow up
Occurrence of Major Cardiovascular Events (MACE) | 52 weeks
  To describe the occurrence of Major Cardiovascular Events (MACE) during the observation period of treatment with BGF, administered as per routine clinical practice Descriptive statistics of the time to first MACE (cardiovascular death, myocardial infarction, or ischemic stroke) occurred during the BGF treatment observation period will be computed by means of a Kaplan-Meier analysis. In case patients do not experience a MACE, they will be considered as censored observations and time until the end of their observation will be calculated. In addition, the count of MACE and the absolute and relative frequency of patients with a MACE will be calculated during the BGF treatment observation period.
Mortality rate | 52 weeks
  To assess the mortality during the observation period of treatment with BGF, administered as per routine clinical practice Descriptive statistics of the time to death occurred during the observation period after BGF treatment start will be computed by means of a Kaplan-Meier analysis. The count of mortality events during the observation period will be reported too.

CONTACTS AND LOCATIONS:
Locations (20):
- Italy (20):
  - Research Site, Acquaviva delle Fonti
  - Research Site, Alessandria
  - Research Site, Ancona
  - Research Site, Avellino
  - Research Site, Brescia
  - Research Site, Brindisi
  - Research Site, Busto Arsizio (Varese)
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Cittadella (Padova)
  - Research Site, Florence
  - Research Site, Foggia
  - Research Site, Lecce
  - Research Site, Napoli
  - Research Site, Passirana (Milano)
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Torino
  - Research Site, Treviso
  - Research Site, Verona

REFERENCES:
- [Background] Gaduzo S, McGovern V, Roberts J, Scullion JE, Singh D. When to use single-inhaler triple therapy in COPD: a practical approach for primary care health care professionals. Int J Chron Obstruct Pulmon Dis. 2019 Feb 13;14:391-401. doi: 10.2147/COPD.S173901. eCollection 2019. PMID 30863039
- [Background] Bourbeau J, Bafadhel M, Barnes NC, Compton C, Di Boscio V, Lipson DA, Jones PW, Martin N, Weiss G, Halpin DMG. Benefit/Risk Profile of Single-Inhaler Triple Therapy in COPD. Int J Chron Obstruct Pulmon Dis. 2021 Mar 1;16:499-517. doi: 10.2147/COPD.S291967. eCollection 2021. PMID 33688176
- [Background] Zheng Y, Zhu J, Liu Y, Lai W, Lin C, Qiu K, Wu J, Yao W. Triple therapy in the management of chronic obstructive pulmonary disease: systematic review and meta-analysis. BMJ. 2018 Nov 6;363:k4388. doi: 10.1136/bmj.k4388. PMID 30401700